CLINICAL TRIAL: NCT03926481
Title: Evaluation of the Healthy Lifestyle Program on Cognitive Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Robert M. Roth, Associate Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D19091
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Obesity
Keywords: weight loss; cognition; sarcopenia; obesity; lifestyle
MeSH Terms: conditions — Obesity; Weight Loss; Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Obesity Only (Experimental): Assess the effect of an intensive lifestyle intervention on cognitive function in adults with obesity who are 65 years and older.
  Interventions: Behavioral: Evaluate Healthy Lifestyle Program on cognitive outcomes
- Sarcopenia and Obesity (Experimental): Assess the effect of an intensive lifestyle intervention on cognitive function in adults with obesity and sarcopenia who are 65 years and older.
  Interventions: Behavioral: Evaluate Healthy Lifestyle Program on cognitive outcomes

INTERVENTIONS:
Behavioral: Evaluate Healthy Lifestyle Program on cognitive outcomes — The healthy lifestyle program will be delivered once a week for 17 weeks as part as regular clinical care. It will include an group classes taught by health coaches and dieticians. These classes will focus on diet, exercise, and behavior modification. We plan 2 cohorts of 15 subjects (n=30). In-person research assistant-led assessments will occur at baseline and 17 weeks.

SUMMARY:
The goal of this study is to conduct a program of pilot research aimed at evaluating the effect of an intensive lifestyle intervention on cognitive functioning in older adults with obesity and or obesity and sarcopenia.

DETAILED DESCRIPTION:
Detailed Description:

The national epidemic of obesity is also affecting older adults, and is associated with an increased risk of disability, nursing home placement and early mortality. The overarching goal of this study is to conduct a program of pilot research aimed at evaluating the effect of a intensive lifestyle intervention on cognitive functioning in order adults with obesity and or obesity and sarcopenia. While some degree of cognitive decline is common during the normal aging process, epidemiological evidence suggests that obesity can promote its acceleration. It is unclear the effect that intensive lifestyle changes could have on cognitive functioning in older adults with obesity.

Study Timeline:

May 2019 to May 2023

Goal: Conduct a study to evaluate the effects that intensive lifestyle program has on cognitive functioning in older adults with obesity and or obesity and sarcopenia.

Participation Duration: Participants will meet weekly for 17 weeks. Cognitive assessments will take place at baseline and 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Age ≥65 years
* Body Composition Body Fat >25% for Men
* Body Composition Body Fat >30% for Women
* Participating in the Dartmouth Hitchcock Weight and Wellness Center (WWC) Healthy Lifestyle Program (HLP)
* Willing and able to give informed consent

Exclusion Criteria:

* Unable to perform measures
* Individuals unwilling/unable to provide consent
* Severe mental or life-threatening illness
* History of bariatric surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Change in grip strength | Baseline and 17 weeks
  Assessed by a Jamar dynamometer. Sensor-based Thera-bands will measure data on strength change. A higher score represents a better outcome.
Change in 5 times Sit-to-Stand (STS) | Baseline and 17 weeks
  STS measures lower limb strength (minimal change 2.3 s). A higher score represents a better outcome.
Change in Six-Minute Walk Test (6MWT) | Baseline and 17 weeks
  A surrogate for cardiovascular fitness that measures distance (normal 400-700m) related to function. A clinically important difference is 50-55m
Change in weight in kg | Baseline and 17 weeks
  Change in weight in kg
Change in body mass index (BMI) in kg/m^2 | Baseline and 17 weeks
  Change in body mass index (BMI) in kg/m^2
Change in subject processing speed | Baseline and 17 weeks
  Single Digit Modalities Test: Measure of cognition/processing speed. Score range 0 to 110. A higher score represents a better outcome.
Change in language function | Baseline and 17 weeks
  Boston Naming Test (BNT) is used to evaluate language function. Score range:0-42; higher score indicates better performance.
Change in subject cognition | Baseline and 17 weeks
  Verbal fluency test is used to evaluate language function. Performance will be identified via the total number of appropriate words responded on each of the task. Higher score indicates better performance.
Change in subject executive function | Baseline and 17 weeks
  Stroop test is used to assess executive function. Higher score indicates better performance. Raw score range: 0-300.
Change in speed processing | Baseline and 17 weeks
  Trail making Test-A&B is used to assess information processing speed. Shorter time indicates better performance.
Change in subject memory | Baseline and 17 weeks
  California Verbal Learning Test II (CVLT-II) Trials 1-5 Total raw score (range: 0-80; higher values represent a better outcome)
Change in Brief Visuospatial Memory Test-Revised (BVMT-R) | Baseline and 17 weeks
  BVMT-R is used to evaluate spatial memory ability. Scores range from 0 to 60, with higher values indicating better performance.
Change from baseline Anxiety Symptoms at 17 weeks | Baseline and 17 weeks
  will be assessed using the Generalized Anxiety Disorder-7 (GAD7). The GAD7 scores range from 5-21, with 5-9 indicating mild, 10-14 moderate, and greater than 15 severe anxiety.
Change from baseline Mood Symptoms at 17 weeks | Baseline and 17 weeks
  Will be assessed using the Patient Healthy Questionnaire (PHQ9). The PHQ9 scores range from 0-27, with lower numbers indicating minimal to no depression and higher numbers indicating severe depression.
Change from baseline Subjective Health Status (PROMIS) at 17 weeks | Baseline and 17 weeks
  Patient Reported Outcomes Measurement Information Systems (PROMIS) Global Short Form. PROMIS is a 10-item instrument capturing physical, mental and social aspects of quality of life having undergone quantitative appraisal and is non-proprietary. Higher score indicated more positive perceptions of overall health.
Change in Behavior Rating Inventory of Executive Function (BRIEF-A) | Baseline and 17 weeks
  Behavior Rating Inventory of Executive Function (BREIF-A) is used to evaluate executive functioning.This questionnaire consist of 75 items on which the patient's symptoms are rated on a 3-point Likert scale. The questionnaire provides a Global Executive Composite score (range 75-225) and two index scores: the Behavioral Regulation Index (range 30-90) and the Metacognitive Index (range 40-120) in addition to nine subscales: Inhibit (range 8-24), Shift (range 6-18), Emotional control (range 10-30), Self-monitor (range 6-18), Initiate (range 8-24), Working memory (range 8-24), Plan/organize (range 10-30), Task monitor (range 6-18) and Organization of materials (range 8-24). Higher scores indicate more executive difficulties.
Change in Prospective and Retrospective Memory Questionnaire (PRMQ) | Baseline and 17 weeks
  PRMQ is a questionnaire about daily memory difficulties. Higher scores represent worse outcomes. Total score ranges from 0-64.

SECONDARY OUTCOMES:
Baseline estimated level of intellectual ability | Baseline
  Test of Premorbid Functioning which results in a total raw score ranging from 0-70, and is normatively scored based on respondents' age resulting in standard scores (mean = 100). Higher values indicate a higher premorbid level of intellect.
Handedness as measured by Edinburgh Handedness Inventory at Baseline | Baseline
  A self report questionnaire assessing the dominance of one's right or left hand in everyday activities.

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Roth, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No